CLINICAL TRIAL: NCT04742673
Title: Maximizing trEatment of Neurological Dysfunction Using INtravenous Guanfacine Study
Acronym: MENDING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christopher G Hughes, Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U11543; 3R01AG053582-05S1 (NIH)
Record Dates: First submitted 2021-01-29; First posted 2021-02-08 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness; Delirium; Cognitive Impairment
MeSH Terms: conditions — Critical Illness; Delirium; Cognitive Dysfunction | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will flow through the trial in the following manner:
  1. Consent in ICU: perform required inclusion/exclusion assessments; discuss study goals, activities, and requirements; obtain informed consent
  2. Pre-randomization phase: twice daily assessments of mental status
  3. Randomize delirious patients: IV guanfacine or placebo
  4. Interventional Trial phase: study drug administration, mental status assessments, safety monitoring
  5. Blood draws: collect blood samples on Interventional Trial Phase days 1 and 2
  6. Follow-up assessments: telephone and online questionnaires at 30, 90, and 180 days after hospital discharge.
  Interventions: Drug: Placebo
- IV Guanfacine (Experimental): Participants will flow through the trial in the following manner:
  1. Consent in ICU: perform required inclusion/exclusion assessments; discuss study goals, activities, and requirements; obtain informed consent
  2. Pre-randomization phase: twice daily assessments of mental status
  3. Randomize delirious patients: IV guanfacine or placebo
  4. Interventional Trial phase: study drug administration, mental status assessments, safety monitoring
  5. Blood draws: collect blood samples on Interventional Trial Phase days 1 and 2
  6. Follow-up assessments: telephone and online questionnaires at 30, 90, and 180 days after hospital discharge.
  Interventions: Drug: Guanfacine

INTERVENTIONS:
Drug: Guanfacine — Patients randomized to the IV Guanfacine arm will receive intravenous guanfacine when they exhibit ICU delirium.
  Arms: IV Guanfacine
Drug: Placebo — Patients randomized to the placebo arm will receive intravenous normal saline when they exhibit ICU delirium.
  Arms: Placebo

SUMMARY:
This proof-of-concept study examines whether the acute brain dysfunction that occurs in critically ill patients is improved by administration of intravenous guanfacine.

DETAILED DESCRIPTION:
Delirium during critical illness is, to date, the primary potentially modifiable risk factor for acquired dementia after critical illness (ADRD). There are, however, no Food and Drug Administration (FDA) approved medications to mitigate delirium. Benzodiazepines are ineffective at reducing the incidence or duration of delirium, and on the contrary, increase the risk. Furthermore, large randomized controlled studies have shown that antipsychotic agents have no effect (vs. placebo) on delirium duration, mechanical ventilation, hospital length of stay, or death. Therefore, current clinical practice guidelines no longer recommend routine use of benzodiazepines or antipsychotics for treatment of delirium. Despite these recommendations, benzodiazepine, antipsychotics, and other drugs are routinely prescribed to critically ill patients due to the urgent clinical need to control delirium symptoms. The alpha-2 agonist dexmedetomidine is the most successful agent for delirium identified to date. However, it is typically administered as a continuous infusion and requires ICU-level monitoring due to hypotension and bradycardia risks. The delirium sparing benefits of dexmedetomidine have been postulated to result from alpha-2 agonist mediated modulation of CNS inflammation, microcirculatory blood flow, and biomimetic sleep.

The alpha-2 agonist guanfacine, an FDA-approved medication for use in hypertension and attention deficit hyperactivity disorder, has a higher selectivity for the alpha-2A receptor in the central nervous system. Thus, delirium sparing benefits may be improved with guanfacine while reducing systemic effects. Further, instead of a continuous infusion, the pharmacokinetic and pharmacodynamic properties of guanfacine favor a twice a day bolus dosing schedule. This Maximizing trEatment of Neurological Dysfunction using INtravenous Guanfacine (MENDING) study will investigate the benefits of intravenous (IV) guanfacine. In this phase II proof-of-concept trial of IV guanfacine vs. placebo for the treatment of critical illness delirium, the following specific aims will be tested in critically ill patients with delirium:

Aim 1: To determine whether IV guanfacine will increase the number of days alive without delirium and coma (DCFDs) over 14 days relative to placebo.

Aim 2: To evaluate whether IV guanfacine twice a day will increase days alive and free of mechanical ventilation (VFDs) and days alive and free of the ICU (IFDs) over 28 days relative to placebo.

Aim 3: To assess whether IV guanfacine can reduce the development of ADRD after critical illness.

Identifying a safe and effective treatment for delirium would have exponential benefits to patients, families, healthcare, and society. This first study of IV guanfacine builds upon extensive research regarding the benefits of alpha-2 agonists for brain dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (≥ 18 years old)
2. requiring admission to an ICU
3. for treatment of respiratory failure (e.g., mechanical ventilation, non-invasive positive pressure ventilation [NIPPV], Extracorporeal Membrane Oxygenation [ECMO], optiflow) and/or for treatment of shock (e.g., vasopressors, ECMO, intra-aortic balloon pump [IABP]).

Exclusion Criteria:

1. allergic to guanfacine, clonidine, or dexmedetomidine
2. on home antipsychotics who, therefore, require continuing antipsychotic administration in the hospital
3. present history of 2nd or 3rd degree heart block, or persistent bradycardia < 50 beats/minute that requires intervention (e.g., atropine, glycopyrrolate). If patient has a pacemaker for bradyarrythmias, then patient does not meet this exclusion criterion and may be enrolled.
4. co-enrolled in another interventional trial examining similar outcomes or in a study that does not allow co-enrollment
5. expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by family or the medical team (e.g., likely withdrawal of life support measures within 24 hours of screening)
6. acute or subacute neurologic deficit that is expected to make the patient incapable of living independently after hospital discharge due to cognitive deficits (e.g., stroke, intracranial hemorrhage, cranial trauma, intracranial malignancy, anoxic brain injury, cerebral edema).
7. dementia or other chronic neurologic disease or disorder that makes the patient incapable of living independently at baseline
8. active substance abuse, psychotic disorder, or homelessness without a secondary contact person (which would make long-term follow-up difficult)
9. blindness or deafness (which would prevent assessment of the study's outcomes)
10. pregnancy or breastfeeding
11. prisoner
12. inability to start informed consent process within 72 hours from the time that all inclusion criteria were met
13. Cardiac surgery within the current hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hughes, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Arnsten AFT, Ishizawa Y, Xie Z. Scientific rationale for the use of alpha2A-adrenoceptor agonists in treating neuroinflammatory cognitive disorders. Mol Psychiatry. 2023 Nov;28(11):4540-4552. doi: 10.1038/s41380-023-02057-4. Epub 2023 Apr 7. PMID 37029295

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | IV Guanfacine
Started | 23 | 23
Completed | 19 | 20
Not Completed | 4 | 3
Not completed — Did not receive any study drug and not included in assessments or results | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | IV Guanfacine | Total
Number analyzed (Participants) | 19 | 20 | 78
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  number analyzed (Participants) | 19 | 20 | 39
  (all) | 65.5 [55.9 to 71.4] | 60.5 [52.5 to 69.6] | 62.3 [54.2 to 71.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 19 | 20 | 39
  Female | 9 | 9 | 18
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  number analyzed (Participants) | 19 | 20 | 39
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 14 | 20 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  number analyzed (Participants) | 19 | 20 | 39
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
SOFA score at ICU admission [Median (Inter-Quartile Range); unit: SOFA score] — Severity of illness at ICU admission as measured by the Sequential Organ Failure Assessment (SOFA) score. This is used to assess the severity of organ dysfunction in critically ill patients, with each organ system (respiratory, cardiovascular, hepatic, coagulation, renal, and central nervous system) receiving a score from 0 (normal) to 4 (most abnormal), resulting in a total score ranging from 0 (normal) to 24 (most abnormal, severe).
  SOFA score
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 10 [7 to 14] | 13.5 [10.75 to 15] | 13 [7.5 to 14.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Alive Without Delirium or Coma
Time Frame: 14 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
days | 7.00 [2.00 to 10.50] | 8.50 [1.75 to 10.00]

2. Secondary Outcome: Days Alive and Free of Mechanical Ventilation
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
days | 22.12 [4.18 to 26.90] | 19.71 [4.45 to 27.00]

3. Secondary Outcome: Days Alive and Free of the Intensive Care Unit
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
days | 19.89 [1.25 to 23.99] | 10.93 [0.00 to 23.01]

4. Secondary Outcome: Cognitive Function
Description: Telephone Montreal Cognitive Assessment has a minimum score of 0 and a maximum score of 22, with higher numbers indicating better cognition. A score of 18 or below is considered a positive screen for at least mild cognitive impairment.
Time Frame: 180 days after randomization
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 10 | 3
Units on a scale | 19.00 [18.50 to 20.50] | 16.00 [15.00 to 16.50]

5. Secondary Outcome: Days Alive and Free of the Hospital
Time Frame: 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
days | 1.00 [0.00 to 7.93] | 0.00 [0.00 to 1.24]

6. Secondary Outcome: Mortality
Time Frame: 90 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
Participants | 6 | 10

7. Other Pre Specified Outcome: Physical Function
Description: Patient-Reported Outcomes Measurement Information System V.1.2-Physical Function 8b is a process that involves using a specific set of 8 questions to assess a patient's self-reported ability to perform physical activities. These questions are designed to measure a person's physical function, focusing on their ability to perform daily activities, including those involving upper and lower extremities, and central body regions. Patients respond to each question on a scale, typically a five-point scale (e.g., 1 = not at all to 5 = completely). The total raw score is then converted to a T-score using a table provided in the PROMIS scoring manual. T-scores are standardized scores with a mean of 50 and a standard deviation of 10, allowing for comparison across individuals and populations. Higher T-scores generally indicate a higher level of physical function.
Time Frame: 180 days after after randomization
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 10 | 3
Units on a scale | 31.9 [27.8 to 39.4] | 36.4 [35.9 to 36.9]

8. Other Pre Specified Outcome: Global Health
Description: Patient-Reported Outcomes Measurement Information System V.1.1-Global is a 10-item questionnaire that measures physical and mental health in patients. The questionnaire uses a T-score metric, where a score of 50 represents the average for the US population with a standard deviation of 10. Higher T-scores indicate better health.
Time Frame: 180 days after after randomization
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 10 | 3
T-score | 37.4 [30.9 to 42.3] | 36.1 [34.2 to 37.9]

9. Other Pre Specified Outcome: Pain Interference
Description: Patient-Reported Outcomes Measurement Information System V.1.0-Pain Interference 8a measures the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. It consists of 8 questions, each with a scale ranging from 1 (Not at all) to 5 (Very much). The score is calculated by summing the responses to all 8 questions, resulting in a raw score range from 8 to 40. This raw score is then converted into a T-score, with a mean of 50 and a standard deviation of 10, and a higher T-score indicating more pain interference.
Time Frame: 180 days after randomization
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 10 | 3
Units on a scale | 59.1 [55.2 to 67.5] | 60.5 [57.3 to 63.7]

10. Other Pre Specified Outcome: Applied Cognition
Description: Patient-Reported Outcomes Measurement Information System V.1.0-Applied Cognition is designed to assess a patient's self-perceived cognitive abilities and concerns in everyday life. The PROMIS measures use a T-score metric with a mean of 50 and a standard deviation of 10, where higher scores indicate better perceived cognitive functioning.
Time Frame: 180 days after randomization
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 10 | 3
Units on a scale | 47.7 [42.5 to 53.5] | 49.6 [47.0 to 52.3]

11. Other Pre Specified Outcome: Sleep
Description: Patient-Reported Outcomes Measurement Information System V.1.0-Sleep Disturbance utilizes a 5-point Likert scale to assess sleep quality, with higher scores indicating greater sleep disturbance. The scale's T-score is a standardized score with a mean of 50 and a standard deviation of 10, with higher scores indicating a greater level of sleep disturbance.
Time Frame: up to 180 days after hospital discharge
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 10 | 3
Units on a scale | 57.0 [48.7 to 64.4] | 52.8 [48.3 to 57.2]

12. Other Pre Specified Outcome: Co-administration of Analgesics
Description: Total opioid dose in fentanyl equivalents
Time Frame: 14 days after randomization
Measure: Median (Inter-Quartile Range); unit: mcg
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
mcg | 4369 [1926 to 8229] | 1883 [638 to 4255]

13. Other Pre Specified Outcome: Hypotension
Description: Refractory systolic blood pressure < 90 mm Hg or Mean arterial blood pressure < 65 mm Hg despite ongoing ICU therapies
Time Frame: 14 days after randomization, while on study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

14. Other Pre Specified Outcome: Bradycardia
Description: Heart rate < 60 beats per minute despite ongoing ICU therapies
Time Frame: 14 days after randomization, while on study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

15. Other Pre Specified Outcome: Mental Status
Description: New, acute neurologic disturbances such as blurred vision, dizziness, weakness, or vertigo
Time Frame: 14 days after randomization, while on study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | IV Guanfacine
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 180 days from randomization
Groups:
- Placebo: Participants will flow through the trial in the following manner:
  1. Consent in ICU: perform required inclusion/exclusion assessments; discuss study goals, activities, and requirements; obtain informed consent
  2. Pre-randomization phase: twice daily assessments of mental status
  3. Randomize delirious patients: IV guanfacine or placebo
  4. Interventional Trial phase: study drug administration, mental status assessments, safety monitoring
  5. Blood draws: collect blood samples on Interventional Trial Phase days 1 and 2
  6. Follow-up assessments: telephone and online questionnaires at 30, 90, and 180 days after hospital discharge.
  Placebo: Patients randomized to the placebo arm will receive intravenous normal saline when they exhibit ICU delirium.
- IV Guanfacine: Participants will flow through the trial in the following manner:
  1. Consent in ICU: perform required inclusion/exclusion assessments; discuss study goals, activities, and requirements; obtain informed consent
  2. Pre-randomization phase: twice daily assessments of mental status
  3. Randomize delirious patients: IV guanfacine or placebo
  4. Interventional Trial phase: study drug administration, mental status assessments, safety monitoring
  5. Blood draws: collect blood samples on Interventional Trial Phase days 1 and 2
  6. Follow-up assessments: telephone and online questionnaires at 30, 90, and 180 days after hospital discharge.
  Guanfacine: Patients randomized to the IV Guanfacine arm will receive intravenous guanfacine when they exhibit ICU delirium.
Arm/Group | Placebo | IV Guanfacine
All-Cause Mortality (participants affected / at risk) | 6/19 | 10/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | IV Guanfacine (N=20)
Fall (Injury, poisoning and procedural complications) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT04742673/Prot_SAP_001.pdf